CLINICAL TRIAL: NCT04559581
Title: Post-marketing Surveillance of Ofev Capsules in Chronic Fibrosing Interstitial Lung Diseases With a Progressive Phenotype in Japan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0402; EUPAS36605 (Registry Identifier: HMA-EMA Catalogues of real-world data sources and studies)
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ofev Capsules: Patients in Japan with Progressive Fibrosing Interstitial Lung Disease (PF-ILD) who were prescribed with Ofev Capsules and were never treated with Ofev Capsules before enrolment, were followed for up to 104 weeks or until discontinuation of administration. The enrollment took place from October 2020 to September 2022.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Ofev Capsules as prescribed by the treating physician
  Other Names: Ofev

SUMMARY:
The primary objective is to evaluate the incidence of adverse drug reactions (focus on hepatic function disorders) of Ofev Capsules under the real world setting in patients with Chronic fibrosing Interstitial Lung Diseases with a progressive phenotype (PF-ILD).

ELIGIBILITY:
Inclusion Criteria:

* Patients in Japan with Chronic fibrosing Interstitial Lung Diseases with a progressive phenotype who are prescribed with Ofev Capsules and have never been treated with Ofev Capsules before enrolment will be included.

Exclusion Criteria:

* Diagnosis of Idiopathic Pulmonary Fibrosis
* Patients with Chronic fibrosing Interstitial Lung Diseases with a progressive phenotype due to systemic scleroderma as the underlying disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-interventional study in patients in Japan with chronic fibrosing ILDs with the progressive phenotype who are prescribed with Ofev and have never been treated with Ofev before; except patients with a diagnosis of idiopathic pulmonary fibrosis or patients with other chronic fibrosing ILDs with the progressive phenotype due to systemic sclerosis as the underlying disease. No limitations are set up on background factors and their concomitant drugs in use of actual medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional study based on newly collected data of patients under routine care to confirm safety of Ofev Capsules (nintedanib) in the real-world setting in Japanese patients with Progressive Fibrosing Interstitial Lung Disease.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
  425 patients were registered, Case Report Forms were collected for 409, and 1 was registered twice, so 408 patients started the treatment.
Period: Overall Study
Arm/Group | Ofev Capsules
Started | 408
Completed | 165
Not Completed | 243
Not completed — Adverse Event | 130
Not completed — Adverse event / Patient's wish | 15
Not completed — Adverse event / Other personal reasons | 2
Not completed — Improved | 2
Not completed — No visit after last visit | 17
Not completed — No visit after last visit / Other personal reasons | 3
Not completed — Other personal reasons | 36
Not completed — Patient's wish | 38

BASELINE CHARACTERISTICS:
Population: Safety set: all patients who didn't have important protocol deviations regarding safety and regulatory issues.
Arm/Group | Ofev Capsules
Number analyzed (Participants) | 408
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 212
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reactions (ADRs)
Description: Incidence of adverse drug reactions (ADRs) is reported as the number of participants with an ADR. An adverse event (AE) was considered to be an ADR if either the physician who reported the AE, or the sponsor, assessed its causal relationship as 'related'.
Time Frame: From first intake of Ofev Capsules prescribed at baseline visit and within 28 days (inclusive) after the last intake of Ofev Capsules, up to approximately 204 weeks.
Population: Safety set: all patients who didn't have important protocol deviations regarding safety and regulatory issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Ofev Capsules
Number analyzed (Participants) | 408
Participants | 246

ADVERSE EVENTS:
Time Frame: From first intake of Ofev Capsules prescribed at baseline visit and within 28 days (inclusive) after the last intake of Ofev Capsules, up to approximately 204 weeks.
Description: Safety set: all patients who didn't have important protocol deviations regarding safety and regulatory issues.
Arm/Group | Ofev Capsules
All-Cause Mortality (participants affected / at risk) | 59/408
Serious Adverse Events (participants affected / at risk) | 139/408
Other Adverse Events (participants affected / at risk) | 192/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofev Capsules (N=408)
Anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 9
Cardiac failure congestive (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 3
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Performance status decreased (General disorders) | 1
Physical deconditioning (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2
Bacterial infection (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 14
Cholangitis infective (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Infectious pleural effusion (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Osteomyelitis chronic (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 13
Pneumonia aspiration (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 10
Pneumonia pseudomonal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Blood pressure decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dermatomyositis (Musculoskeletal and connective tissue disorders) | 1
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Nephritis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 67
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Microscopic polyangiitis (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral circulatory failure (Vascular disorders) | 1
Vascular pain (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofev Capsules (N=408)
Diarrhoea (Gastrointestinal disorders) | 123
Nausea (Gastrointestinal disorders) | 36
Hepatic function abnormal (Hepatobiliary disorders) | 32
Liver disorder (Hepatobiliary disorders) | 25
Decreased appetite (Metabolism and nutrition disorders) | 26

LIMITATIONS AND CAVEATS:
Due to the nature of a single cohort observational study, there are issues that may impose limitations, in particular on the validity of the assessment based on the study data, such as selection bias, loss to follow up, channeling bias, and information and recall bias. Thus, comparisons and causal conclusions cannot be made, except for the investigator reported drug-related adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04559581/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04559581/SAP_001.pdf